CLINICAL TRIAL: NCT00605423
Title: A Single Masked, Randomized Comparison of the Safety and Efficacy of 0.2 and 0.5 µg/Day Fluocinolone Acetonide/Medidur™ in Patients With Exudative Age Related Macular Degeneration Who Have Received Lucentis™
Brief Title: The MAP Study: Fluocinolone Acetonide (FA)/Medidur (TM) for Age Related Macular Degeneration (AMD) Pilot
Acronym: MAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Alimera Sciences (Industry); pSiVida Limited (Industry)
Responsible Party: Principal Investigator, Peter A Campochiaro, MD, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA 00012714
Record Dates: First submitted 2008-01-17; First posted 2008-01-31 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD; Almera; Steroid; Macular; ARMD
MeSH Terms: conditions — Macular Degeneration | interventions — Fluocinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Dose 0.2 ug/day Medidur implant
  Interventions: Drug: Fluocinolone Acetonide/Medidur
- 2 (Active Comparator): Dose 0.5 ug/day Medidur implant
  Interventions: Drug: Fluocinolone Acetonide/Medidur

INTERVENTIONS:
Drug: Fluocinolone Acetonide/Medidur — 0.2 ug/day implant
  Arms: 1
Drug: Fluocinolone Acetonide/Medidur — 0.5 ug/day implant
  Arms: 2

SUMMARY:
Treatment of exudative age-related macular degeneration has been significantly improved by the advent of Lucentis™( which provides improved vision rather than simply stabilization) is common; however, monthly injections may be required to maintain this effect. It is hypothesized that sustained release fluocinolone acetonide will allow maintenance of the improved vision with fewer Lucentis injections.

DETAILED DESCRIPTION:
Treatment of exudative age-related macular degeneration has been significantly improved by the advent of Lucentis™( which provides improved vision rather than simply stabilization) is common; however, monthly injections may be required to maintain this effect. The use of the glucocorticoids such as triamcinolone acetonide as adjunct treatment for exudative age-related macular degeneration has been reported to enhance the efficacy of photodynamic therapy with Visudyne® (verteporphin for injection). It is hypothesized that sustained release fluocinolone acetonide will allow maintenance of the improved vision with fewer Lucentis injections. This study is a pilot phase 2b study to test this hypothesis. The safety assessments will continue through 36 months.This study will compare the safety 2 doses of FA/Medidur in conjunction with Lucentis (as needed) in patients with neovascular AMD who have have been treated with Lucentis for at least 6 months and have reached a plateau.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 or greater
* Treated with intraocular injections of Lucentis for at least 6 months and have reached a plateau, defined as 2 consecutive visits (4-6 weeks apart) with no improvement in VA (worse or within one line better) or center subfield thickening (worse or within 30 um better).
* Best Corrected Visual Acuity 20/320 or better in the study eye

Exclusion Criteria:

* Pregnant, lactating females or females of child bearing potential (unless using reliable contraception, i.e. double barrier, surgical sterilization, oral contraceptives, Norplant , intrauterine device (IUD).
* Glaucoma or ocular hypertension (defined as IOP > 21 mmHg or concurrent therapy at screening with IOP-lowering agents) in the study eye
* Laser or photodynamic therapy within 12 weeks of screening
* Any ocular surgery in the study eye within 12 weeks of screening
* Yag capsulotomy in the study eye within 15 days of screening
* Treatment with intravitreal, subtenon, or periocular steroid or anti-VEGF therapy other than Lucentis within 6 months prior to enrollment (e.g., triamcinolone injection, Avastin, Macugen.) Systemic treatment with Avastin is also not allowed within 6 months prior to screening or at any time during the study.
* Any change in systemic steroid therapy within 3 months of screening
* Retinal or choroidal neovascularization due to ocular conditions other than AMD.
* Any active viral, fungal or bacterial disease of the cornea or conjunctiva or any history of a potentially recurrent infection which could be activated by treatment with a steroid, (e.g., ocular herpes simplex virus).
* Known or suspected hypersensitivity to any of the ingredients of Lucentis, the investigational product or to other corticosteroids.
* History of vitrectomy in the study eye
* History of uncontrolled IOP elevation with steroid use that did not respond to topical therapy
* History or presence of any disease or condition (malignancy) that in the investigator's opinion would preclude study treatment or follow-up
* Any lens opacity which impairs visualization of the posterior pole
* Participation in another clinical trial within 12 weeks before the screening visit or during the study
* Subjects who are a poor medical risk because of other systemic diseases or active uncontrolled infections.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Campochiaro, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluocinolone Acetonide: 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur implant
- Fluocinolone Acetonide: 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur implant
Period: Overall Study
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluocinolone Acetonide: 0.2 ug/Day Implant: Dose 0.2 ug/day Medidur implant
  Fluocinolone Acetonide/Medidur : 0.2 ug/day implant
- Fluocinolone Acetonide: 0.5 ug/Day Implant: Dose 0.5 ug/day Medidur implant
  Fluocinolone Acetonide/Medidur : 0.5 ug/day implant
- Total: Total of all reporting groups
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (5.3) | 75.9 (3.9) | 75.5 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Visual Acuity
Description: Visual acuity is measured using ETDRS charts at 4 meters.
Time Frame: 6 mos
Measure: Mean (Standard Deviation); unit: ETDRS letters
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 4 | 2
ETDRS letters | 1.8 (5.19) | 1.0 (8.49)

2. Secondary Outcome: Number of Patients Developing Cataracts
Time Frame: 6 mos
Measure: Number; unit: participants
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 4 | 2
participants | 4 | 2

3. Secondary Outcome: Change in IOP From Baseline
Description: IOP stands for intra ocular pressure
Time Frame: 6 mos
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Number analyzed (Participants) | 4 | 2
mmHg | 1.30 (5.81) | 2.65 (1.91)

ADVERSE EVENTS:
Arm/Group | Fluocinolone Acetonide: 0.2 ug/Day Implant | Fluocinolone Acetonide: 0.5 ug/Day Implant
Serious Adverse Events (participants affected / at risk) | 4/4 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=4) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=2)
Cataract Operation (Surgical and medical procedures) | 4 (4) | 1 (1)
Cataract Operation Complication (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluocinolone Acetonide: 0.2 ug/Day Implant (N=4) | Fluocinolone Acetonide: 0.5 ug/Day Implant (N=2)
Cataract (Eye disorders) | 3 (3) | 2 (2) — Study Eye
Cataract Subcapsular (Eye disorders) | 1 (3) | 0 (0) — Study Eye
Contrast Media Reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraocular Pressure Increased (Investigations) | 1 (1) | 1 (1) — Study Eye
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cataract Operation Complication (Surgical and medical procedures) | 1 (1) | 0 (0) — Study Eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days